CLINICAL TRIAL: NCT04924192
Title: A Clinical Study of TQB3616 Capsules Combined With Anlotinib Hydrochloride Capsules or Standard Chemotherapy Second-line and Above in the Treatment of Advanced Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB3616-ALTN-II-01
Record Dates: First submitted 2021-06-10; First posted 2021-06-11 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Advanced Lung Carcinoma
MeSH Terms: interventions — Irinotecan; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB3616 capsules+Anlotinib hydrochloride capsules (Experimental): TQB3616 capsules 120/150/180mg orally on an empty stomach, once a day for 21 consective days as a treatment cycle;Anlotinib hydrochloride capsules 12mg, once a day for 2 consecutive weeks and stop for 1 week.
  Interventions: Drug: TQB3616 capsules; Drug: Anlotinib Hydrochloride capsules
- TQB3616 capsules +Irinotecan Hydrochloride for Injection (Experimental): TQB3616 capsules 120/150/180mg orally on an empty stomach, once a day for 28 consecutive days as a treatment cycle. Irinotecan Hydrochloride Injection 100 mg/m2 intravenous infusion on D1、D8 and D15, a total of 4-6 cycles.
  Interventions: Drug: TQB3616 capsules; Drug: Irinotecan Hydrochloride for Injection

INTERVENTIONS:
Drug: TQB3616 capsules — A CDK4/6 kinase inhibitor
Drug: Anlotinib Hydrochloride capsules — A multi-target receptor tyrosine kinase inhibitor
  Arms: TQB3616 capsules+Anlotinib hydrochloride capsules
Drug: Irinotecan Hydrochloride for Injection — An inhibitor of DNA topoisomerase Ⅰ
  Arms: TQB3616 capsules +Irinotecan Hydrochloride for Injection

SUMMARY:
This is an open, multi-cohort, exploratory phase II study on the safety and efficacy of TQB3616 combined with Anlotinib hydrochloride capsules or standard chemotherapy in the treatment of advanced lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with pathologically proven small cell lung cancer(SCLC) or/and locally advanced ( Stage ⅢB/ ⅢC), metastatic or recurrent (Stage IV) non small cell lung cancer(NSCLC).
2. Cohort 1: Subjects with SCLC who had previously received at least one chemotherapy containing platinum or got disease progression during chemoradiotherapy or after the last treatment.
3. Cohort 2: Subjects with locally advanced, metastatic/relapsed NSCLC who had previously received only one PD (L) 1 inhibitor alone or in combination with platinum-based chemotherapy.
4. Subjects with measurable lesions as defined by RECIST 1.1.
5. Aged ≥ 18 years ; Eastern Cooperative Oncology Group (ECOG) score: 0 ~ 1; Expected survival ≥ 3 months.
6. Laboratory indicators meet the requirements.
7. Non-pregnant or non-breastfeeding women; Negative pregnancy subjects.
8. Subjects voluntarily joined the study and signed the informed consent form.

Exclusion Criteria:

1. Subjects who received prior therapy with anlotinib hydrochloride capsules.
2. Cohort 2: Subjects with epidermal growth factor receptor(EGFR) mutation and anaplastic lymphoma kinase(ALK) translocation.
3. Subjects with central squamous cell carcinoma with a risk of hemoptysis.
4. Subjects who have developed or is currently suffering from other malignancies within 5 years, with the exception of cured skin basal cell carcinoma and cervical carcinoma in situ.
5. Subjects who have brain metastases with symptoms or control of symptoms for less than 2 months.
6. Subjects with difficulty taking oral medication.
7. Subjects with uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage.
8. Subjects with spinal cord compression who have failed to be cured or relieved by surgery and or radiotherapy.
9. Subjects who have received chemotherapy, radiotherapy or other experimental anticancer therapy within 4 weeks prior to the first dose of the drug.
10. Subjects who have not recovered to ≤ CTCAE Grade 1 (excluding alopecia) due to the adverse event of prior therapy.
11. Subjects with significant surgery or significant traumatic injury within 28 days before randomization.
12. Subjects with arterial/venous thrombosis within 6 months.
13. Subjects with a history of psychotropic substance abuse who cannot be withdrawn or have mental disorders.
14. Subjects with any severe and/or uncontrolled disease.
15. Subjects whose large vessels are involved by tumor from imaging (CT or MRI).
16. Subjects who have hemoptysis and maximum daily hemoptysis ≥ 2.5ml within 1 month before the first dose.
17. Subjects with other factors that might cause the study to be terminated halfway per the judgement of the investigator.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-05-23 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 96 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 96 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Disease control rate（DCR） | up to 96 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Response (DOR) | up to 120 weeks
  The time when the participants first achieved CR or PR to disease progression or death from any cause.
6-month progression-free survival rate | up to 96 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
6-month and 12-month overall survival rate | up to 96 weeks
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The Second Affiliated Hospital of PLA Air Force Military Medical University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdou, Sichuan
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan